CLINICAL TRIAL: NCT02083562
Title: Plasma Biomarkers for the Prediction of Bronchopulmonary Dysplasia and Volumetric Capnography for Severity Assessment of Lung Disease in Preterm Infants
Brief Title: Biomarkers and Volumetric Capnography in BPD
Acronym: BPD-2014
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BPD-2014_UKBB
Record Dates: First submitted 2014-02-25; First posted 2014-03-11 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia, preterm infant
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the association of biomarkers on day 7 of life with the development of bronchopulmonary dysplasia in very preterm infants. Additionally a short lung function test at 36 weeks postmenstrual age (PMA) will be performed to investigate whether certain capnographic indices are able to reflect the degree of lung disease.

Protocol was amended (under others: additional enrollment of 70 subjects).

DETAILED DESCRIPTION:
This is a two-centre prospective cohort study in very preterm infants born below 32 0/7 weeks PMA and hospitalised in the neonatal intensive care units at the University Children's Hospital Basel and the Inselspital Berne during two years. After informed consent a sample of 0.5 mL ethylenediaminetetraacetic acid (EDTA) full blood will be taken on day 7 of life (+/- 2 days) during routine blood sampling. The biomarkers which are planned to measure include the C-terminal portion of the proendothelin-1 precursor (CT-proendothelin (proET)-1) and other plasma biomarkers of respiratory distress. At 36 weeks PMA, lung function testing will be performed during quiet unsedated sleep in supine position approximately 30 minutes post feeding. After placement of a facemask, tidal breathing will be recorded at the bedside using a commercially available ultrasonic flow meter (Spiroson, Exhalyzer D, Ecomedics, CH) according to American Thoracic Society (ATS) and European Respiratory Society (ERS) standards of infant lung function testing. Different capnographic indices will be calculated to investigate if they reflect the degree of lung disease at 36 weeks PMA.

ELIGIBILITY:
Inclusion Criteria:

* parental consent, born below 32 weeks PMA

Exclusion Criteria:

* No parental consent, major life-threatening anomalies (cardiac defects, primary pulmonary malformations etc.)

Ages: 5 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born below 32 weeks PMA and admitted to the neonatal intensive care units in Basel and Berne, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
association of plasma biomarker levels (pro-endothelin-1 precursor and other markers of respiratory distress) with the duration of supplemental oxygen dependancy in infancy | Assessment at 36 weeks PMA or until the end of supplemental oxygen dependancy assessed up to 12 months
association of capnographic indices with the duration of supplemental oxygen dependancy | 36 weeks PMA or until the end of supplemental oxygen dependancy assessed up to 12 months
  Capnographic indices include expired carbon dioxide volume per breath, slopes of phase II (SII) and slopes of phase III (SIII) of the capnogram.

SECONDARY OUTCOMES:
several definitions of BPD | 36 weeks PMA
duration of respiratory support | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
death | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
sepsis | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
necrotizing enterocolitis (NEC) | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
retinopathy of prematurity (ROP) | until completion of retinal vascularization or up to 6 months, whichever came first
intraventricular hemorrhage (IVH) | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
patent ductus arteriosus | participants will be followed for the duration of hospital stay, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland P Neumann, MD, Principal Investigator — Department of Neonatology, University Children's Hospital Basel, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Department of Neonatology, University Children's Hospital Basel, Basel
  - Department of Neonatology, Inselpital Berne, Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Neumann RP, Gerull R, Zannin E, Fouzas S, Schulzke SM. Volumetric Capnography at 36 Weeks Postmenstrual Age and Bronchopulmonary Dysplasia in Very Preterm Infants. J Pediatr. 2022 Feb;241:97-102.e2. doi: 10.1016/j.jpeds.2021.10.019. Epub 2021 Oct 24. PMID 34687691